CLINICAL TRIAL: NCT01182779
Title: Randomised Trial of Proton vs. Carbon Ion Radiation Therapy in Patients With Chordoma of the Skull Base -Clinical Phase III Study-
Brief Title: Trial of Proton Versus Carbon Ion Radiation Therapy in Patients With Chordoma of the Skull Base
Acronym: HIT-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Juergen Debus, MD PhD, Dept. of Radiation Oncology, INF 400, 69120 Heidelberg, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIT-1
Record Dates: First submitted 2010-07-26; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-07

CONDITIONS: Chordoma; Tumor; Treatment
Keywords: base of skull chordoma; radiation; carbon ions; protons
MeSH Terms: conditions — Chordoma; Neoplasms | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Arm A (carbon ion therapy):
  Total dose to the PTV2 - 45 Gy E in 3 Gy E /d, 4-6 days a week, 15 fractions Total dose to the PTV1 - 63 Gy E ± 5%, further 5-7 fractions a 3 Gy E.
  Interventions: Radiation: Carbon ion
- B (Active Comparator): Arm B (proton therapy):
  Total dose to the PTV2 - 50 to 56 Gy E in 2 Gy E /d, 4-6 days a week, 28 fractions Total dose to the PTV1 - 72 Gy E ± 5%, further 6-9 fractions a 2 Gy E.
  Interventions: Radiation: Protons

INTERVENTIONS:
Radiation: Carbon ion — Arm A (carbon ion therapy):
  Total dose to the PTV2 - 45 Gy E in 3 Gy E /d, 4-6 days a week, 15 fractions Total dose to the PTV1 - 63 Gy E ± 5%, further 5-7 fractions a 3 Gy E.
  Arms: A
Radiation: Protons — Arm B (proton therapy):
  Total dose to the PTV2 - 50 to 56 Gy E in 2 Gy E /d, 4-6 days a week, 28 fractions Total dose to the PTV1 - 72 Gy E ± 5%, further 6-9 fractions a 2 Gy E.
  Arms: B

SUMMARY:
This study is a prospective randomised clinical phase III trial. The primary objective of this study is to evaluate, if the innovative therapy (carbon ion irradiation) in chordomas is superior to the standard proton treatment with respect to the local-progression free survival (LPFS).

DETAILED DESCRIPTION:
The study is a prospective randomised clinical phase III trial. The trial will be carried out at Heidelberger Ionenstrahl-Therapie (HIT) centre as monocentric trial.

Proton therapy is the gold standard in the treatment of skull base chordomas. However, high-LET beams such as carbon ions theoretically offer biologic advantages by enhanced biologic effectiveness in slow-growing tumors. Up until now it was impossible to compare two different particle therapies, i.e. proton and carbon ion therapy directly with each other. The aim of this study is to find out, whether the biological advantages of carbon ion therapy mentioned above can also be clinically confirmed.

Patients with skull base chordoma will be randomised to either proton or carbon ion radiation therapy. As a standard, patients will undergo non-invasive, rigid immobilization and target volume delineation will be carried out based on CT and MRI data. The biologically isoeffective target dose to the PTV in carbon ion treatment (accelerated dose) will be 63 Gy E ± 5% and 72 Gy E ± 5% (standard dose) in proton therapy respectively. Local-progression free survival (LPFS) will be analysed as primary end point. Toxicity and survival are the secondary end points. Also matters of interest are patterns of recurrence, prognostic factors and plan quality.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score ≥60%
* Age >18 years and <80 years
* Informed consent signed by the patient
* Histological confirmation of chordoma with infiltration of the skull base.

Exclusion Criteria:

* Inability to understand the aims of the study, no informed consent
* Prior RT of skull base region
* Other malignancies with disease-free interval < 5 years (excepting pre- cancerous lesions)
* Participation in another trial
* Pregnancy
* Simultaneous CHT or Immunotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
local-progression free survival (LPFS) | 8-years
  The primary objective of this study is to evaluate, if the innovative therapy (carbon ion irradiation) in chordomas is superior to the standard proton treatment with respect to the LPFS defined as time from the randomisation to observed local reccurrence or death from any cause in the absence of documented local disease progression. Lo-cal recurrence defined as MRT or CT - morphological tumor progress in the former irradiated region. A 10% increase in the LPFS is considered clinically relevant as-suming that the LPFS rate for the proton therapy is 70%.

SECONDARY OUTCOMES:
Survival | 8-years
  Assessment of overall survival, progression free and metastasis free survival.
Local control and patterns of recurrence | 8 years
  Local recurrences will be confirmed radiologically and histologically whenever possible. At least two medical doctors (radiation oncologist and/or radiologist) will be required to judge of the recurrence.
Toxicity | 8 years
  Acute and late toxicity will be analysed due to Common Terminology Criteria for Adverse Events: CTCAE V4.0 for acute reaction and RTOG/EORTC for late effects.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD PhD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Munzenrider JE, Liebsch NJ. Proton therapy for tumors of the skull base. Strahlenther Onkol. 1999 Jun;175 Suppl 2:57-63. doi: 10.1007/BF03038890. PMID 10394399
- [Background] Ares C, Hug EB, Lomax AJ, Bolsi A, Timmermann B, Rutz HP, Schuller JC, Pedroni E, Goitein G. Effectiveness and safety of spot scanning proton radiation therapy for chordomas and chondrosarcomas of the skull base: first long-term report. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1111-8. doi: 10.1016/j.ijrobp.2008.12.055. Epub 2009 Apr 20. PMID 19386442
- [Background] Hug EB. Review of skull base chordomas: prognostic factors and long-term results of proton-beam radiotherapy. Neurosurg Focus. 2001 Mar 15;10(3):E11. doi: 10.3171/foc.2001.10.3.12. PMID 16734403
- [Background] Hug EB, Slater JD. Proton radiation therapy for chordomas and chondrosarcomas of the skull base. Neurosurg Clin N Am. 2000 Oct;11(4):627-38. PMID 11082173
- [Background] Weber DC, Rutz HP, Pedroni ES, Bolsi A, Timmermann B, Verwey J, Lomax AJ, Goitein G. Results of spot-scanning proton radiation therapy for chordoma and chondrosarcoma of the skull base: the Paul Scherrer Institut experience. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):401-9. doi: 10.1016/j.ijrobp.2005.02.023. PMID 16168833
- [Background] Schulz-Ertner D, Karger CP, Feuerhake A, Nikoghosyan A, Combs SE, Jakel O, Edler L, Scholz M, Debus J. Effectiveness of carbon ion radiotherapy in the treatment of skull-base chordomas. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):449-57. doi: 10.1016/j.ijrobp.2006.12.059. Epub 2007 Mar 23. PMID 17363188
- [Background] Mizoe JE, Hasegawa A, Takagi R, Bessho H, Onda T, Tsujii H. Carbon ion radiotherapy for skull base chordoma. Skull Base. 2009 May;19(3):219-24. doi: 10.1055/s-0028-1114295. PMID 19881902
- [Derived] Nikoghosyan AV, Karapanagiotou-Schenkel I, Munter MW, Jensen AD, Combs SE, Debus J. Randomised trial of proton vs. carbon ion radiation therapy in patients with chordoma of the skull base, clinical phase III study HIT-1-Study. BMC Cancer. 2010 Nov 5;10:607. doi: 10.1186/1471-2407-10-607. PMID 21054824